CLINICAL TRIAL: NCT05045079
Title: Tricuspid Regurgitation Due to Atrial Fibrillation - Impact of Rhythm Control and Early Surgery (TR-ES Study)
Brief Title: Rhythm Control and Potential Early Surgery for Tricuspid Regurgitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yogesh Reddy, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-000537
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Severe Tricuspid Valve Regurgitation (Disorder)
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe tricuspid regurgitation due to atrial fibrillation (Other): Subjects will receive standard of care procedure right heart catheterization with a inferior vena caval (IVC) occlusion maneuver.
  Interventions: Procedure: Inferior Vena Caval (IVC) Occlusion maneuver

INTERVENTIONS:
Procedure: Inferior Vena Caval (IVC) Occlusion maneuver — During standard of care right heart catheterization (RHC), a second catheter will be inserted next to the catheter that was placed for the RHC in the jugular vein or femoral vein to assess the degree of pericardial restraint from the severe tricuspid regurgitation that may increase left sided filling pressures.

SUMMARY:
The purpose of this study is to understand the clinical impact of non-surgical and surgical treatment in atrial fibrillation induced tricuspid regurgitation (AFTR).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Moderate-severe or severe TR while in atrial fibrillation.
* Ambulatory (not wheelchair/scooter dependent).

Exclusion Criteria:

* Systolic pulmonary artery pressure>70 mmHg with a fixed pulmonary vascular resistance >7 Wood units by catheterization.
* Ejection fraction <40%.
* Obstructive hypertrophic cardiomyopathy.
* Constrictive pericarditis or tamponade.
* Active myocarditis.
* Complex congenital heart disease.
* Other valve disease requiring surgical intervention.
* Terminal illness (other than HF) with expected survival of less than 1 year.
* Pregnancy or breastfeeding mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Change in KCCQ QOL scores | Baseline, 6 months
  The KC Cardiomyopathy Questionnaire (0-100 scale) assess subject perception of heart failure limitation on their life; scale of extremely limited, quite a bit limited, moderately limited, slightly limited, not at all limited, limited for other reasons or did not do the activity.

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Reddy, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials